CLINICAL TRIAL: NCT01336413
Title: Neuroactive Steroids and TBI in OEF/OIF Veterans
Brief Title: Neuroactive Steroids and Traumatic Brain Injury (TBI) in OEF/OIF Veterans
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B4603-I; NCT01327131 (obsolete NCT alias)
Record Dates: First submitted 2011-04-13; First posted 2011-04-15 (Estimated); Results first posted 2017-10-20 (Actual); Last update posted 2019-07-12 (Actual); Status verified 2017-09

CONDITIONS: Brain Injuries, Traumatic
Keywords: brain injuries, traumatic; pregnenolone; Veteran; OEF/OIF; neurosteroid; allopregnanolone
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Pregnenolone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 (Active Comparator): Pregnenolone
  Interventions: Drug: Pregnenolone
- Arm 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pregnenolone — Pregnenolone 50 mg BID x 14 DAYS, followed by Pregnenolone 150 mg BID x 14 DAYS, followed by Pregnenolone 250 mg BID x thereafter for the remainder of the 8-week trial
  Arms: Arm 1
Drug: Placebo — Same as active comparator, except placebo dispensed.
  Arms: Arm 2

SUMMARY:
Purpose: Mild traumatic brain injury (TBI) is extremely common among Operation Enduring Freedom/Operation Iraqi Freedom (OEF/OIF) era Veterans. Mild TBI is frequently accompanied by post-traumatic stress disorder (PTSD) and depression symptoms, co-occurring disorders that contribute to increased disability and decreased quality of life. Neuroactive steroids (NS) represent promising pharmacological candidates for intervention for these diverse symptom domains, since a number of these molecules demonstrate pronounced neuroprotective and neurotrophic properties. The NS pregnenolone (PREG) is a logical therapeutic option, since it enhances learning and memory and also increases myelination in rodent models. Further, decreases in PREG have been associated with depressive symptoms, and PREG is also metabolized to allopregnanolone (ALLO), an anxiolytic downstream NS that is decreased in PTSD. ALLO also enhances neurogenesis in rodents. The investigators thus propose an randomized controlled trial (RCT) in OEF/OIF era Veterans with mild TBI.

Methodology: The design of this study will be randomized, placebo-controlled, double-blind. Trial duration will be 10 weeks, consisting of a 2-week placebo lead-in period for all subjects, followed by 8 weeks of treatment with either pregnenolone or placebo. The primary cognitive outcome measure will be executive functioning (as assessed by the Tower of London test), and the primary behavioral outcome measure will be PTSD Cluster D symptoms (as assessed by the Clinician-Administered PTSD Scale, CAPS). The investigators will also determine if PREG administration in OEF/OIF Veterans with mild TBI increases downstream ALLO and/or other GABAergic NS levels, and the investigators will identify the specific metabolism profile of PREG following eight weeks of treatment with this neurosteroid.

Anticipated Findings: The investigators hypothesize that treatment with PREG in OEF/OIF era Veterans with mild TBI will significantly improve executive functioning compared to the placebo condition. The investigators also predict that treatment with PREG will decrease Cluster D PTSD symptoms compared to treatment with placebo.

DETAILED DESCRIPTION:
Purpose: Mild traumatic brain injury (TBI) is extremely common among OEF/OIF (Operation Enduring Freedom/Operation Iraqi Freedom) era Veterans. Mild TBI is frequently accompanied by post-traumatic stress disorder (PTSD) and depression symptoms, co-occurring disorders that contribute to increased disability and decreased quality of life. Neuroactive steroids (NS) represent promising pharmacological candidates for intervention for these diverse symptom domains, since a number of these molecules demonstrate pronounced neuroprotective and neurotrophic properties. The NS pregnenolone (PREG) is a logical therapeutic option, since it enhances learning and memory and also increases myelination in rodent models. Further, decreases in PREG have been associated with depressive symptoms, and PREG is also metabolized to allopregnanolone (ALLO), an anxiolytic downstream NS that is decreased in PTSD. ALLO also enhances neurogenesis in rodents. The investigators thus propose an RCT in OEF/OIF era Veterans with mild TBI.

Methodology: The design of this study will be randomized, placebo-controlled, double-blind. Trial duration will be 10 weeks, consisting of a 2-week placebo lead-in period for all subjects, followed by 8 weeks of treatment with either pregnenolone or placebo. The primary cognitive outcome measure will be executive functioning (as assessed by the Tower of London test), and the primary behavioral outcome measure will be PTSD Cluster D symptoms (as assessed by the Clinician-Administered PTSD Scale, CAPS). The investigators will also determine if PREG administration in OEF/OIF Veterans with mild TBI increases downstream ALLO and/or other GABAergic NS levels, and the investigators will identify the specific metabolism profile of PREG following eight weeks of treatment with this neurosteroid. A subset of patients will also receive pre/post neuroimaging (functional magnetic resonance imaging [fMRI], diffusion tensor imaging [DTI], and quantitative susceptibility mapping/susceptibility tensor imaging [QSM/STI]).

Anticipated Findings: The investigators hypothesize that treatment with PREG in OEF/OIF era Veterans with mild TBI will significantly improve executive functioning compared to the placebo condition. The investigators also predict that treatment with PREG will decrease Cluster D PTSD symptoms compared to treatment with placebo.

ELIGIBILITY:
Inclusion Criteria:

* 21-55 years of age, any ethnic group, either sex
* History of mild TBI since 2001
* The investigators will adhere to the operational definition of mild TBI suggested by the World Health Organization Task Force (Holm et al 2005), with the exception of Glasgow Coma Scale score criteria (not available for these subjects): a.) One or more of the following: confusion or disorientation, loss of consciousness for 30 minutes or less, post-traumatic amnesia for less than 24 hours, and/or other transient neurological abnormalities such as focal signs, seizure, and intracranial lesion not requiring surgery; Glasgow Coma Scale (GCS) score of 13-15 after 30 minutes post-injury or later upon presentation for health care (GCS unavailable). This WHO diagnostic definition of mild TBI is also consistent with the CDC Report to Congress on Mild TBI in the United States, September 2003 (specifically, altered consciousness attributable to the head injury [=transient confusion, disorientation or impaired consciousness] or self reported loss of consciousness lasting 30 minutes or less).
* Ability to participate fully in the informed consent process.
* No anticipated need to alter psychiatric medications for the 10-week duration of the study. Since this study is adjunctive to treatment-as-usual, patients will not be tapered from any psychiatric medications they may be receiving at enrollment.
* No changes in psychotropic or behavioral interventions during the study or in the 4 weeks prior to study enrollment.

Exclusion Criteria:

* For this pilot study, the investigators will diverge slightly from the above WHO definition of mild TBI and exclude patients who report a history of seizures for this investigation. Although no seizures have been reported to the FDA in relationship to pregnenolone use, pregnenolone could theoretically influence seizure threshold if metabolized to its sulfated derivative, which demonstrates negative modulatory actions at GABAA receptors. Since the preliminary data suggest that pregnenolone administration increases the GABAergic neuroactive steroid allopregnanolone five-fold, however, and since allopregnanolone demonstrates marked anticonvulsant activity in a number of animal seizure models, this theoretical risk may be small or non-existent.
* Subjects with current suicidal or homicidal ideation necessitating clinical intervention or representing an imminent concern.
* Concomitant medications for medical conditions will be addressed on a case-by-case base and determined if exclusionary.
* Current DSM-IV diagnosis of bipolar disorder, schizophrenia or other psychotic disorder, or cognitive disorder due to a general medical condition other than TBI.
* Female patients who are pregnant or breast-feeding.
* Known allergy to study medication.
* Substance dependence or abuse (other than nicotine dependence), as determined by MINI assessment.
* Serious unstable medical illness. History of cerebrovascular accident, prostate, uterine or breast cancer.
* Use of oral contraceptives or other hormonal supplementation such as estrogen [although early studies suggested no effects on menstrual cycle, alterations in downstream metabolites of pregnenolone could theoretically impact efficacy of oral contraceptives and estrogen replacement].

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 53 (Actual)
Dates: Start 2013-10; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christine Marx, MD MA, Principal Investigator — Durham VA Medical Center, Durham, NC
Locations (1):
- Durham VA Medical Center, Durham, NC, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pregnenolone | Placebo
Started | 27 | 26
Completed | 26 | 18
Not Completed | 1 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pregnenolone | Placebo | Total
Number analyzed (Participants) | 27 | 26 | 53
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.74 (5.40) | 35.04 (6.75) | 33.87 (6.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 26 | 25 | 51
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 6 | 9
  White | 19 | 18 | 37
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 27 | 26 | 53

OUTCOME MEASURES:

1. Primary Outcome: CAPS (Cluster D Symptoms) - PRIMARY BEHAVIORAL OUTCOME MEASURE
Description: The CAPS-IV criterion D is defined by persistent symptoms of increasing arousal (not present before the trauma), indicated by at least two of the following: difficulty falling or staying asleep, irritability or outbursts of anger, difficulty concentrating, hyper-vigilance, and exaggerated startle response There are two scales, frequency and intensity. Frequency scores range from 0 = "none of the time" to 4 = "most or all of the time" and intensity scores range from 0 = "none" to 4 = "extreme." Severity scores are calculated from the sum of frequency and intensity scores. Five items are included in criterion D, thus the range of severity scores is 0-45. Higher scores are indicative of more symptoms.
Time Frame: Baseline, 4 Weeks, and 8 Weeks
Population: 3 subjects in Arm 1, and 1 subject in Arm 2, withdrew prior to the final visit of the study
Measure: Mean (Standard Error); unit: Score
Arm/Group | Pregnenolone | Placebo
Number analyzed (Participants) | 26 | 18
Score
  Baseline | 13.88 (1.51) | 12.89 (2.07)
  4 Weeks | 11.23 (1.63) | 10.89 (2.33)
  8 Weeks: number analyzed (Participants) | 23 | 17
  8 Weeks | 9.13 (1.46) | 12.24 (2.32)

2. Primary Outcome: Tower of London (Subscale Test of BAC) - PRIMARY COGNITIVE OUTCOME MEASURE
Description: Subscale test asking subjects to determine the minimum number of moves that will be required to make convert one image of colored balls on pegs into a second different image. The test administers 20 items/images, with 2 additional items if all of the first 20 are answered correctly. Thus, scores range from 0-22, with lower scores representing greater impairment. Raw scores are converted to z scores that generally range from -3 to 3, with lower scores again representing greater impairment.
Time Frame: Baseline, 4 Weeks, and 8 Weeks
Population: 3 subjects in Arm 1, and 1 subject in Arm 2, withdrew prior to the final visit of the study.
Measure: Mean (Standard Error); unit: z Score
Arm/Group | Pregnenolone | Placebo
Number analyzed (Participants) | 26 | 18
z Score
  Baseline | 0.23 (0.14) | -0.17 (0.24)
  4 Weeks | 0.36 (0.15) | 0.14 (0.22)
  8 Weeks: number analyzed (Participants) | 23 | 17
  8 Weeks | 0.20 (0.17) | 0.43 (0.21)

3. Secondary Outcome: Beck Depression Inventory-II (BDI-II)
Description: 21-item, self-report rating inventory that measures characteristic attitudes and symptoms of depression. Scores range from 0 (no depression) to 63 (severe depression).
Time Frame: Baseline, 4 Weeks, and 8 Weeks
Population: 3 subjects in Arm 1, and 1 subject in Arm 2, withdrew prior to the final visit of the study.
Measure: Mean (Standard Error); unit: Total Score
Arm/Group | Pregnenolone | Placebo
Number analyzed (Participants) | 26 | 18
Total Score
  Baseline | 11.27 (1.15) | 10.56 (2.30)
  4 Weeks | 8.42 (1.24) | 8.44 (1.89)
  8 Weeks: number analyzed (Participants) | 23 | 17
  8 Weeks | 7.30 (0.87) | 8.88 (2.05)

4. Secondary Outcome: BAC Composite
Description: Composite z scores (allowing comparison from week 2 to week 10) to assess cognitive changes. The BAC includes brief assessments of executive functions, verbal fluency, attention, verbal memory, working memory and motor speed. z scores are calculated from composite scores. Higher z scores are indicative of better cognitive performance, lower z scores are indicative of lower cognitive performance. Range of z scores anticipated to be between -3 and 3.
Time Frame: Baseline, 4 Weeks, and 8 Weeks
Population: 3 subjects in Arm 1, and 1 subject in Arm 2, withdrew prior to the final visit of the study.
Measure: Mean (Standard Error); unit: Composite z Score
Arm/Group | Pregnenolone | Placebo
Number analyzed (Participants) | 26 | 18
Composite z Score
  Baseline | -0.14 (0.22) | -0.59 (0.26)
  4 Weeks | 0.26 (0.20) | -0.10 (0.29)
  8 Weeks: number analyzed (Participants) | 23 | 17
  8 Weeks | 0.18 (0.26) | 0.17 (0.28)

5. Secondary Outcome: CAPS Total Scores
Description: Mean scores in posttraumatic stress disorder symptoms. Scores may range from 0 (no symptoms) to 136 (severe symptoms; score of 136 is based on the first 17 CAPS items administered). A reduced CAPS score indicates a reduction in (improvement) PTSD symptoms, while and increase in CAPS score indicates an increase (worsening) in PTSD symptoms.
Time Frame: Baseline, 4 Weeks, and 8 Weeks
Population: 3 subjects in Arm 1, and 1 subject in Arm 2, withdrew prior to the final visit of the study.
Measure: Mean (Standard Error); unit: Total Score
Arm/Group | Pregnenolone | Placebo
Number analyzed (Participants) | 26 | 18
Total Score
  Baseline | 32.04 (4.02) | 33.33 (5.72)
  4 Weeks | 23.65 (3.52) | 26.22 (6.24)
  8 Weeks: number analyzed (Participants) | 23 | 17
  8 Weeks | 22.83 (4.04) | 27.47 (6.52)

6. Secondary Outcome: Connor-Davidson Resilience Scale (CD-RISC)
Description: The CD-RISC was developed and tested as (i) a measure of degree of resilience, (ii) as a predictor of outcome to treatment with medication or psychotherapy, stress management and resilience-building, (iii) as a marker of progress during treatment, and (iv) as a marker of biological changes in the brain. The scale comprises 25 items, each rated on a 5-point scale (0-4) for a total range of 0-100, with higher scores reflecting greater resilience.
Time Frame: Baseline, 4 Weeks, and 8 Weeks
Population: 3 subjects in Arm 1, and 1 subject in Arm 2, withdrew prior to the final visit of the study.
Measure: Mean (Standard Error); unit: Total Score
Arm/Group | Pregnenolone | Placebo
Number analyzed (Participants) | 26 | 18
Total Score
  Baseline | 70.19 (2.38) | 69.06 (4.42)
  4 Weeks | 71.73 (2.45) | 72.22 (3.87)
  8 Weeks: number analyzed (Participants) | 23 | 17
  8 Weeks | 72.13 (2.62) | 73.11 (4.00)

7. Other Pre Specified Outcome: Functional Magnetic Resonance Imaging (Exploratory Neuroimaging Outcome)
Description: Functional Magnetic Resonance Imaging (fMRI) to assess possible functional brain changes related to attention and emotion circuits associated with the intervention. The dependent measure is the BOLD (fMRI) response to images of faces expressing neutral emotions and fearful emotions.
Time Frame: 10 weeks
Measure: Mean (Standard Error); unit: BOLD percent signal change in vmPFC
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 11 | 6
BOLD percent signal change in vmPFC
  pre-treatment neutral condition | -3.598 (1.978) | 5.288 (2.678)
  pre-treatment fear condition | 0.767 (2.506) | -3.208 (3.393)
  post-treatment neutral condition | -0.781 (2.018) | -6.917 (2.732)
  post-treatment fear condition | -5.05 (3.112) | 5.472 (4.214)

8. Other Pre Specified Outcome: Diffusion Tensor Imaging (Exploratory Neuroimaging Outcome)
Description: Diffusion Tensor Imaging (DTI) to assess possible white matter brain changes associated with intervention.
Time Frame: 10 weeks
Measure: Mean (Standard Error); unit: fractional anisotropy index units
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 13 | 7
fractional anisotropy index units
  corpus callosum pre-treatment | 0.5518 (0.007) | 0.5477 (0.0088)
  corpus callosum post-treatment | 0.5416 (0.0083) | 0.5432 (0.0093)
  anterior corona radiata pre-treatment | 0.5211 (0.0082) | 0.5151 (0.0103)
  anterior corona radiata post-treatment | 0.5072 (0.0089) | 0.5118 (0.0106)
  anterior limb of internal capsule pre-treatment | 0.4750 (0.0055) | 0.4732 (0.0080)
  anterior limb of internal capsule post-treatment | 0.4670 (0.0073) | 0.4694 (0.0081)
  cerebral peduncle pre-treatment | 0.5920 (0.0054) | 0.5812 (0.0050)
  cerebral peduncle post-treatment | 0.5784 (0.0089) | 0.5797 (0.0111)
  cingulum cingulate gyrus pre-treatment | 0.5729 (0.0081) | 0.5706 (0.0079)
  cingulum cingulate gyrus post-treatment | 0.5598 (0.0098) | 0.5663 (0.0113)
  cingulum hippocampus pre-treatment | 0.4379 (0.0070) | 0.4227 (0.0095)
  cingulum hippocampus post-treatment | 0.4152 (0.0105) | 0.4210 (0.0136)
  corpus callous splenium pre-treatment | 0.4042 (0.0116) | 0.4151 (0.0213)
  corpus callous splenium post-treatment | 0.3759 (0.0177) | 0.3893 (0.0304)
  corticospinal tract pre-treatment | 0.5979 (0.0068) | 0.5987 (0.0112)
  corticospinal tract post-treatment | 0.5888 (0.0093) | 0.5891 (0.0106)
  external capsule pre-treatment | 0.4269 (0.0141) | 0.4407 (0.0095)
  external capsule post-treatment | 0.4236 (0.0080) | 0.4329 (0.0099)
  fornix column pre-treatment | 0.3944 (0.0039) | 0.3925 (0.0082)
  fornix column post-treatment | 0.3782 (0.0081) | 0.3821 (0.0112)
  Inferior cerebellar peduncle pre-treatment | 0.4347 (0.0073) | 0.4295 (0.0106)
  Inferior cerebellar peduncle post-treatment | 0.4302 (0.0078) | 0.4254 (0.0094)
  Medial Lemniscus pre-treatment | 0.5100 (0.0075) | 0.5017 (0.0094)
  Medial Lemniscus post-treatment | 0.4961 (0.0108) | 0.4933 (0.0142)
  Posterior corona radiata pre-treatment | 0.5071 (0.0048) | 0.5021 (0.0096)
  Posterior corona radiata post-treatment | 0.4897 (0.0100) | 0.4943 (0.0124)
  Posterior limbs of internal capsule pre-treatment | 0.5448 (0.0057) | 0.5319 (0.0103)
  Posterior limbs of internal capsule post-treatment | 0.5252 (0.0103) | 0.5264 (0.0118)
  posterior thalamic radiation pre-treatment | 0.5819 (0.0057) | 0.5695 (0.0085)
  posterior thalamic radiation post-treatment | 0.5687 (0.0094) | 0.5622 (0.0093)
  retrolenticular part of internal capsule pre-treat | 0.5780 (0.0076) | 0.5569 (0.0115)
  retrolenticular part of internal capsule posttreat | 0.5582 (0.0106) | 0.5511 (0.0118)
  Sagittal Stratum pre-treatment | 0.5316 (0.0063) | 0.5136 (0.0076)
  Sagittal Stratum post-treatment | 0.5146 (0.0112) | 0.5104 (0.0114)
  Superior cerebellar peduncle pre-treatment | 0.5267 (0.0058) | 0.5291 (0.0119)
  Superior cerebellar peduncle post-treatment | 0.5066 (0.0112) | 0.5170 (0.0146)
  Superior Corona radiata pre-treatment | 0.5009 (0.0058) | 0.5091 (0.0132)
  Superior Corona radiata post-treatment | 0.4835 (0.0100) | 0.5020 (0.0165)
  Superior fronto-occipital fasciulus pre-treatment | 0.4571 (0.0062) | 0.4574 (0.0122)
  Superior fronto-occipital fasciulus post-treatment | 0.4453 (0.0085) | 0.4540 (0.0126)
  Superior longitudinal fascicles pre-treatment | 0.4557 (0.0072) | 0.4464 (0.0139)
  Superior longitudinal fascicles post-treatment | 0.4445 (0.0087) | 0.4432 (0.0121)
  Tapetum pre-treatment | 0.3758 (0.0092) | 0.3751 (0.0086)
  Tapetum post-treatment | 0.3645 (0.0098) | 0.3727 (0.0082)
  Uncinate fasciculus pre-treatment | 0.3997 (0.0063) | 0.4147 (0.0096)
  Uncinate fasciculus post-treatment | 1.3893 (0.0072) | 0.4105 (0.0105)

9. Other Pre Specified Outcome: Quantitative Susceptibility Mapping/Susceptibility Tensor Imaging (Exploratory Neuroimaging Outcome)
Description: Quantitative Susceptibility Mapping/Susceptibility Tensor Imaging (QSM/STI) to assess possible myelin brain changes related to the intervention.
Time Frame: 10 weeks
Measure: Mean (Standard Error); unit: magnetic susceptibility ratio
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 14 | 10
magnetic susceptibility ratio
  red nucleus pre-treatment | -0.0236 (0.0057) | -0.0253 (0.0038)
  red nucleus post-treatment | -0.0246 (0.0031) | -0.0312 (0.0053)
  substantia nigra pre-treatment | -0.0376 (0.0085) | -0.0399 (0.0047)
  substantia nigra post-treatment | -0.0456 (0.0034) | -0.0481 (0.0048)
  pulvinar pre-treatment | -0.0421 (0.0035) | -0.0395 (0.0055)
  pulvinar post-treatment | -0.0391 (00035) | -0.0427 (0.0078)
  dentate nucleus pre-treamtment | -0.0071 (0.0046) | -0.0059 (0.0056)
  dentate nucleus post-treatment | -0.0116 (0.0033) | -0.0092 (0.0066)
  corpus callosum genu pre-treatment | 0.0093 (0.0015) | 0.0045 (0.0034)
  corpus callosum genu post-treatment | 0.0096 (0.0027) | -0.0011 (0.0031)
  corpus callosum body pre-treatment | 0.0049 (0.0020) | 0.0063 (0.0019)
  corpus callosum body post-treatment | 0.0036 (0.0018) | 0.0059 (0.0046)
  anterior corona radiata pre-treatment | 0.0142 (0.0025) | 0.0060 (0.0012)
  anterior corona radiata post-treatment | 0.0084 (0.0024) | 0.0025 (0.0015)
  anterior limb internal capsule pre-treatment | 0.0094 (0.0028) | 0.0047 (0.0034)
  anterior limb internal capsule post-treatment | 0.0099 (0.0022) | 0.0036 (0.0026)
  cerebral peduncle pre-treatment | 0.0141 (0.0040) | 0.134 (0.004)
  cerebral peduncle post-treatment | 0.0133 (0.0033) | 0.0036 (0.0034)
  cingulate cingulum pre-treatment | 0.0016 (0.0011) | 0.0021 (0.0019)
  cingulate cingulum post-treatment | 0.0017 (0.0008) | 0.0037 (0.002)
  cingulum hippocampus pre-treatment | -0.00630 (0.0024) | -0.0042 (0.0024)
  cingulum hippocampus post-treatment | -0.0041 (0.0008) | -0.0042 (0.0031)
  corpus callosum splenium pre-treatment | 0.0149 (0.0011) | 0.0146 (0.0014)
  corpus callosum splenium post-treatment | 0.0103 (0.0018) | 0.0098 (0.0007)
  cortico-spinal pre-treatment | 0.0209 (0.0023) | 0.0168 (0.0012)
  cortico-spinal post-treatment | 0.0178 (0.0008) | 0.0166 (0.0018)
  external capsule pre-treatment | 0.0002 (0.006) | 0.0054 (0.0009)
  external capsule post-treatment | 0.0048 (0.0011) | 0.0074 (0.0011)
  fornix column body pre-treatment | -0.0118 (0.0048) | -0.0171 (0.0028)
  fornix column body post-treatment | -0.011 (0.0041) | -0.0221 (0.0014)
  interior cerebellar peduncle pre-treatment | 0.0120 (0.0018) | 0.0118 (0.0011)
  interior cerebellar peduncle post-treatment | 0.0088 (0.0009) | 0.0119 (0.0015)
  medial lemniscus pre-treatment | 0.0236 (0.0015) | 0.0197 (0.0014)
  medial lemniscus post-treatment | 0.0212 (0.0018) | 0.0217 (0.0022)
  posterior corona radiate pre-treatment | 0.0133 (0.0014) | 0.0121 (0.0011)
  posterior corona radiate post-treatment | 0.144 (0.0009) | 0.0131 (0.0007)
  posterior limb internal capsule pre-treatment | 0.0270 (0.0026) | 0.0267 (0.0018)
  posterior limb internal capsule post-treatment | 0.0292 (0.0014) | 0.0267 (0.0017)
  posterior thalamic radiation pre-treatment | 0.0184 (0.0015) | 0.0181 (0.0009)
  posterior thalamic radiation post-treatment | 0.0201 (0.001) | 0.0199 (0.0013)
  retrolenticular internal capsule pre-treatment | 0.0018 (0.0058) | 0.0039 (0.0022)
  retrolenticular internal capsule post-treatment | 0.0077 (0.0009) | 0.0043 (0.0016)
  sagittal stratum pre-treatment | 0.0145 (0.0016) | 0.0138 (0.0025)
  sagittal stratum post-treatment | 0.0148 (0.0010) | 0.0160 (0.0011)
  superior cerebellar peduncle pre-treatment | 0.0049 (0.0016) | 0.0076 (0.0028)
  superior cerebellar peduncle post-treatment | 0.0055 (0.0019) | 0.0082 (0.0025)
  superior corona radiata pre-treatment | 0.0086 (0.0014) | 0.0090 (0.0008)
  superior corona radiata post-treatment | 0.0096 (0.0006) | 0.0098 (0.0007)
  superior fronto-occipital fasciculus pre-treatment | 0.0033 (0.0017) | 0.0061 (0.0018)
  superior fronto-occipital fasciculus post-treatmt | 0.0021 (0.0016) | 0.0064 (0.0018)
  superior longitudinal fasciculus pre-treatment | 0.0024 (0.0028) | 0.0047 (0.0007)
  superior longitudinal fasciculus post-treatment | 0.0049 (0.0005) | 0.0055 (0.0011)
  tapetum pre-treatment | 0.0031 (0.0023) | 0.0023 (0.0016)
  tapetum post-treatment | 0.0015 (0.0017) | 0.0045 (0.0016)
  uncinate fasciculus pre-treatment | 0.0219 (0.0038) | 0.0268 (0.0021)
  uncinate fasciculus post-treatment | 0.0250 (0.0016) | 0.0260 (0.0031)

ADVERSE EVENTS:
Arm/Group | Pregnenolone | Placebo
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/26
Other Adverse Events (participants affected / at risk) | 22/27 | 13/26
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pregnenolone (N=27) | Placebo (N=26)
Headache (General disorders) | 15 (30) | 10 (26)
Dermatological (Skin and subcutaneous tissue disorders) | 6 (8) | 1 (1)
Restlessness (General disorders) | 5 (6) | 3 (6)
Insomnia (General disorders) | 2 (5) | 2 (3)
Irritabilty (General disorders) | 3 (3) | 2 (3)
Dry Mouth (General disorders) | 3 (3) | 4 (9)
Diarrhea (Gastrointestinal disorders) | 2 (3) | 0 (0)
Akathisia (General disorders) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (2) | 1 (1)
Nasal Congestion (General disorders) | 2 (2) | 1 (1)
Nausea (General disorders) | 1 (1) | 3 (4)
Malaise (General disorders) | 1 (1) | 0 (0)
Tremor (General disorders) | 1 (1) | 1 (1)
Decreased Appetite (General disorders) | 1 (1) | 0 (0)
Decreased Motor Activity (General disorders) | 1 (1) | 0 (0)
Drowsiness (General disorders) | 1 (1) | 1 (1)
Increased Motor Activity (General disorders) | 1 (1) | 0 (0)
Joint Pain/Stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle Pain/Stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Paresthesia (General disorders) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Blurred Vision (Eye disorders) | 0 (0) | 1 (1)
Cramps (General disorders) | 0 (0) | 1 (1)
Increased Appetite (General disorders) | 0 (0) | 1 (2)
Sweating (General disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes